CLINICAL TRIAL: NCT01259661
Title: Physical Activity and Metabolic Risk Factors in Postmenopausal Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Jen-Chen Tsai, School of Nursing, Taipei Medical University
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 99070
Record Dates: First submitted 2010-12-07; First posted 2010-12-14 (Estimated); Last update posted 2010-12-14 (Estimated); Status verified 2010-12

CONDITIONS: Postmenopausal Women
Keywords: physical activity; metabolic syndrome; postmenopausal women; exercise training
MeSH Terms: conditions — Motor Activity; Metabolic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental Group (Experimental)
  Interventions: Other: A longitudinal intervention
- Control Group (Active Comparator)
  Interventions: Other: A longitudinal intervention

INTERVENTIONS:
Other: A longitudinal intervention — In our longitudinal intervention study, all eligible subjects will undergo a physical examination by a physician to rule out obvious secondary causes of hypertension and contraindications to exercise. Randomization will be performed by random member generation. The exercise participants will attend three sessions per week at the facility during the study period. Training intensity is initially set at heart rate equivalent to 60% and progress to 80% of each subject's maximal heart rate reserve for 30 min/day with a frequency of 3 days/wk. Facility-based exercise sessions will consist of treadmill walking.

SUMMARY:
Hormonal changes associated with menopause, chronological aging, and lifestyle, especially physical inactivity, may increase the risk of metabolic syndrome in postmenopausal women. Women exhibiting "the metabolic syndrome" have multiple coronary artery disease risk factors, including insulin resistance, hyperlipidemia, and hypertension. This study will be conducted to test the hypotheses: (1) physical activity and physical fitness levels may have effects on individual risk factors of the metabolic syndrome in postmenopausal women; (2) endurance exercise training may have a favorable effect on components of the metabolic risk variables in these women.

In this study, the associations among physical activity (including daily energy expenditure and energy expenditure from moderate to vigorous activity), cardiopulmonary fitness level, and metabolic risk profile of the women will be assessed. The investigators will perform a randomized trial to compare the effects of moderate-intensity aerobic exercise training regimens on metabolic risk factors. Postmenopausal women who exhibit at least one risk factor for metabolic syndrome will be randomized in the exercise group or control groups. Metabolic risk factors (e.g., body mass index, waist-to-hip ratio, glucose, insulin, blood pressure, lipid profile and adiponectin level) will be measured at baseline, and 12 weeks of the study. Differences from baseline to follow-up will be calculated and compared across groups.

Results of this study may help health care providers providing advice to postmenopausal women for life style changes to reduce risk of insulin resistance, coronary heart disease, and diabetes.

ELIGIBILITY:
Inclusion Criteria:

* have one or more metabolic risk variables as defined by the ATP III (2001)
* age between 35 and 64 years
* absence of known heart disease
* resting BP: 130 < SBP < 160 and 85 < DBP < 100
* currently physical inactive (< 30 min of physical activity per week)

Exclusion Criteria:

* None of the participants has a diagnosis of type 2 diabetes, physical illness or disabilities that will limit daily physical activities.

Ages: 35 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2010-10; Primary Completion 2011-10 (Estimated); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
Postmenopausal women's daily energy expenditure | 12 week

CONTACTS AND LOCATIONS:
Overall Officials: Jen-Chen Tsai, Principal Investigator — Taipei Medical University
Locations (1):
- Taipei Medical University WanFang Hospital, Taipei, Taiwan